CLINICAL TRIAL: NCT05036148
Title: Malignant Hyperthermia in Czech Republic: Description of the Biggest Slavonic Group of Patients Investigated for Risk of Malignant Hyperthermia (MH): Retrospective MH Registry Analysis
Brief Title: Malignant Hyperthermia in Czech Republic: Description of the Biggest Slavonic Group of Patients Investigated for Risk of Malignant Hyperthermia
Acronym: MHCZECH
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: KDAR FN Brno MH
Record Dates: First submitted 2021-07-27; First posted 2021-09-05 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Malignant Hyperthermia
Keywords: Malignant Hyperthermia
MeSH Terms: conditions — Malignant Hyperthermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients indicated for MH screening: Patients referred to MH center for MH diagnostic
  Interventions: Other: Data analysis

INTERVENTIONS:
Other: Data analysis — MH registry data will be screened for MH positive diagnosis

SUMMARY:
The Academic centre for Malignant Hyperthermia of Masaryk University (ACMHMU) was established in 2021 in Brno, Czech Republic and consists of four academic departments of Medical Faculty of Masaryk University in two tertiary university hospitals, University Hospital Brno and St. Anne Faculty Hospital. These departments collaborated and operated since 2002 and since 2019 is Brno one of the of centre of EMHG (www.emhg.org). Aim of this study was to describe the Czech and Slovak (CZ-SK) cohort of MHS patients, the biggest Slavonic MHS cohort known by now, and to fill the knowledge gap about the Slavonic population in perspective of MH.

DETAILED DESCRIPTION:
We evaluated every referral to the MH centre since 2002 then. IVCT results, clinical data, personal and family history and molecular genetic data, have been recorded in an electronic medical record. Potential MHS patients, probands, were investigated according to the European Malignant Hyperthermia Group (EMHG) recommendations using IVCT and/or RYR1 and CACNA1S sequence variant screening. Each proband is a representative of one unrelated family. As the diagnostic guidelines were changing in the time, so was our diagnostic algorithm with the development of new knowledge and methods.

Originally before 2015, for each proband or the nearest relative in case that the index case could not be tested, MH must be confirmed/excluded by IVCT. Only with a positive IVCT positive result (MHS, MHEh, MHEc), genetic diagnosis was originated.

iIn 2015, a new EMHG guideline for the diagnosis of MH was issued and significantly moved the DNA diagnosis of MH to the forefront and we started to use genetic testing as a first diagnostic step. Not finding the diagnostic variant does not exclude MH susceptibility and IVCT needs to follow for final diagnosis. IVCT has been providing according to the best practise and EMGH guidelines.

So far, the genetic diagnosis of MH in the Czech Republic has been in several stages - starting with standard scoring of 33 most common causal diagnostic variants of the RYR1 gene by using multiplex ligation-dependent probe amplification (MLPA) (SALSA MLPA probemix P281-A3/P282-A3 RYR1, MRC Holand). In case of a negative result, direct sequence analysis of the RYR1 and CACNA1S gene sections followed, where the remaining causal diagnostic variants occur. Since 2021 MLPA and direct sequencing of hot spots regions of RYR1 and CACNA1S was routinely replaced by next-generation sequencing (NGS) at the level of a panel of genes associated with neuromuscular diseases (including RYR1, CACNA1S and STAC3).

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated to MH center for MH diagnostic

Exclusion Criteria:

* conditions clearly not related to MH, e.g. neuromuscular diseases
* syndromes without MH risk; anaesthetic complications without MH symptoms, e.g. prolongated awakening due to deficit of cholinesterase
* probands with missing data
* probands with yet not closed MH diagnostic process (waiting for genetics or IVCT, myopatic patients without MH diagnostic variant where the IVCT was not recommended because of its invasivity)
* non-compliant probands, who refused the diagnostic process.

Ages: 1 Month to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient indiaceted to MH centre for MH diagnostic
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
prevalence of MH in our cohort of patients | 20 years retrospectively
  Data registry will be screened for positive MH results

SECONDARY OUTCOMES:
prevalence of occurrence diagnostic variants in MHS group of patients. | 20 years retrospectively
  Data registry will be screened for different MH gene variants
prevalence of each found diagnostic variant in our Czech-and-Slovak cohort of patients. | 20 years retrospectively
  Data registry will be screened for each found diagnostic variant in our Czech-and-Slovak cohort of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., Study Chair — Department of paediatric anaesthesia and intensive care
Locations (1):
- Brno University Hospital - Academic Centre for Malignant Hyperthermia of Masaryk University Brno, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided